CLINICAL TRIAL: NCT01367080
Title: Clinical Trials to Compare the Pharmacokinetics Profile of Etravil®(Amitriptyline Hydrochloride) Tablet 10mg and Etravil®(Amitriptyline Hydrochloride) Tablet 25mg After a Single Oral Administration in Healthy Male Volunteers
Brief Title: A Study to Compare the Pharmacokinetic Profiles of Etravil® Tablet 10mg and Etravil® Tablet 25mg
Acronym: DWETR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Collaborators: Chonbuk National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DWETR-I-1
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Depression; Depressive State; Enuresis
Keywords: depression
MeSH Terms: conditions — Depression; Enuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A Group (Experimental): 1. 1st administration - DWETR10
  2. 2nd administration - DWETR25
  Interventions: Drug: DWETR10; Drug: DWETR25
- B Group (Experimental): 1. 1st administration - DWETR25
  2. 2nd administration - DWETR10
  Interventions: Drug: DWETR10; Drug: DWETR25

INTERVENTIONS:
Drug: DWETR10 — Amitriptyline hydrochloride 10mg(DWETR10) single dose
  Other Names: Etravil 10mg
Drug: DWETR25 — Amitriptyline hydrochloride 25mg(DWETR25) single dose
  Other Names: Etravil 25mg

SUMMARY:
To evaluate the pharmacokinetics of single oral dose of Amitriptyline hydrochloride film-coated tablet 10mg & 25mg

DETAILED DESCRIPTION:
Randomized, Single dose, 2-way crossover, Open Study to compare the pharmacokinetics profile of Etravil®(Amitriptyline Hydrochloride) Tablet 10mg and Etravil®(Amitriptyline Hydrochloride) Tablet 25mg after a single oral administration in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* a healthy adult male within the range of 19 to 50 years old at the time of screening
* one with weight of more than 55kg, in the range of IBW 20%

  * Ideal Body Weight(IBW)(kg)={height(cm)-100}*0.9
* one who understood completely about this study after the detailed explanation is given, decided to volunteer and gave written informed consent to participate in study in compliance with the requirement of the entire protocol.

Exclusion Criteria:

* one with clinically significant disease in liver, kidney, nerve system, respiratory system, endocrine system, blood, tumor, urinary system, cardiovascular system, mental disease or with medical history
* one with glaucoma
* one with disorders of micturition include benign prostatic hyperplasia
* one with gastrointestinal disease or with gastrointestinal surgical history which can affect the absorption of the investigational drug.
* one who is allergic or has clinically significant allergic history to the study drug, components or tricyclic antidepressants(TCA)
* one who shows the following result in vital sign: hypotension(systolic pressure ≤ 100mmHg or diastolic pressure ≤ 65mmHg) or hypertension(systolic pressure ≥ 150mmHg or diastolic pressure ≥ 95mmHg)
* one who has drug abuse history
* one who has taken any prescribed drugs, herbal agents or crude drugs within 2 weeks before study drug administration, or who has taken any over-the-counter (OTC) drugs or vitamins (Investigators will determine his eligibility by considering the effect of the drug on his safety or pharmacokinetic results in case other inclusion/exclusion criteria is satisfied.)
* one who has participated in other clinical study within 2 months before study drug administration
* one who donated whole blood within 2 months or component blood within 1 month or who are donated within 1 month before the treatment
* one who drank Over 21 units/week of alcohol(1 unit = 10g of pure alcohol) or subjects who would not be able to stop drinking alcohol during the hospitalization
* one who are heavy smoker more than 10 cigarettes/day within 3 months prior to screening or subjects who would not be able to stop smoking during the hospitalization
* one who had a beverage containing caffeine, drank alcohol, or smoked within 48hrs before the hospitalization or who had a beverage containing grapefruits during the hospitalization
* one with clinically significant observations considered as unsuitable based on medical judgment by investigators

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, MD, PhD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital., Jeonju, Jeollabuk-do, South Korea

REFERENCES:
- [Derived] Nam Y, Lim CH, Lee HS, Chung SJ, Chung YH, Shin YK, Kim MG, Sohn UD, Kim HC, Jeong JH. Single-dose, randomized, open-label, 2-way crossover study of the pharmacokinetics of amitriptyline hydrochloride 10- and 25-mg tablet in healthy male Korean volunteers. Clin Ther. 2015 Feb 1;37(2):302-10. doi: 10.1016/j.clinthera.2014.09.010. Epub 2014 Oct 11. PMID 25308868

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from a specialty clinic at a hospital, Korea between July 2011 and August 2011
Pre-assignment Details: 15 participants recruited ; 12 screened, 3 excluded (2 did not meet inclusion criteria and 1 refused participation)
Groups:
- A Group: Etravil tablet 10mg once daily in first intervention period and Etravil tablet 25mg once daily in second intervention period (10days washout period, Intervention period : 1day)
- B Group: Etravil tablet 25mg once daily in first intervention period and Etravil tablet 10mg once daily in second intervention period (10days washout period, Intervention period : 1day)
Period: 1st Administration
Arm/Group | A Group | B Group
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: 2nd Administration
Arm/Group | A Group | B Group
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A Group | B Group | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.2 (2.1) | 21.2 (2.1) | 21.7 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: AUClast and AUCinf
Description: Area Under the Plasma concentration-time curve from time Zero to Infinity(AUCinf) and Area Under the Plasma concentration-time curve from time Zero to last time(AUClast) of Amitryptiline in plasma
Time Frame: Up to 72 hours
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Etravil 10mg Group: Amitryptiline Hydrochloride 10mg administration Group
- Etravil 25mg Group: Amitryptiline hydrochloride 25mg administration Group
Arm/Group | Etravil 10mg Group | Etravil 25mg Group
Number analyzed (Participants) | 12 | 12
ng*hr/mL
  AUClast | 91.35 (25.88) | 260.68 (111.57)
  AUCinf | 109.74 (37.80) | 296.87 (124.99)

2. Secondary Outcome: Cmax
Description: Maximum Concentration(Cmax) of amitryptyline in plasma
Time Frame: Up to 72 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Etravil 10mg Group | Etravil 25mg Group
Number analyzed (Participants) | 12 | 12
ng/mL | 5.96 (1.40) | 17.69 (5.27)

3. Secondary Outcome: Tmax
Description: Time for Maximum Concentration(Tmax) of Amitryptyline in Plasma
Time Frame: Up to 72 hours
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Etravil 10mg Group | Etravil 25mg Group
Number analyzed (Participants) | 12 | 12
hour | 3.50 (0.90) | 3.13 (0.61)

4. Secondary Outcome: t1/2
Description: Terminal half-time(t1/2) of Amitryptyline in Plasma
Time Frame: Up to 72 hours
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Etravil 10mg Group | Etravil 25mg Group
Number analyzed (Participants) | 12 | 12
hour | 26.47 (5.64) | 24.79 (3.22)

ADVERSE EVENTS:
Time Frame: About a month
Groups:
- Etravil 10mg Group: Amitryptyline hydrochloride 10mg administration Group
- Etravil 25mg Group: Amitryptyline hydrochloride 25mg administration Group
Arm/Group | Etravil 10mg Group | Etravil 25mg Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etravil 10mg Group (N=12) | Etravil 25mg Group (N=12)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
When collecting blood samples, few subjects were drawn blood later than that stated in protocol for about 1 ~ 2 minutes where results may not be effected.

One of the subjects came in late for Post-study visit for about 4~6 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No